CLINICAL TRIAL: NCT04982874
Title: Bioequivalence Study of Furosemide in Indonesian Healthy Volunteers
Brief Title: Bioequivalence Study of Furosemide 40 mg Tablet in 24 Indonesian Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Kimia Farma (Persero) Tbk (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 447/STD/PML/2019
Record Dates: First submitted 2021-07-18; First posted 2021-07-29 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-01

CONDITIONS: Drug Use
Keywords: bioequivalence; furosemide; Indonesian healthy volunteers
MeSH Terms: interventions — Furosemide; Tablets

STUDY DESIGN:
Intervention Model Description: randomized, single blind, single dose, 2-period, cross-over design with one week washout period between each treatment in 24 healthy volunteers beneath fasting condition
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide 40 mg tablet (Experimental): volunteers received Furosemide 40 mg tablet with 240 mL of water
  Interventions: Drug: Furosemide 40 mg
- Lasix® 40 mg Tablet (Active Comparator): volunteers received Lasix® 40 mg tablet with 240 mL of water
  Interventions: Drug: Lasix® 40 mg Tablet

INTERVENTIONS:
Drug: Furosemide 40 mg — Administered with 240 mL of water
  Arms: Furosemide 40 mg tablet
Drug: Lasix® 40 mg Tablet — Administered with 240 mL of water
  Other Names: Furosemide 40 mg
  Arms: Lasix® 40 mg Tablet

SUMMARY:
The purpose of this research was to investigate whether Furosemide 40 mg tablet manufactured by PT. Kimia Farma Tbk was bioequivalent to its reference drug and Lasix® 40 mg Tablet manufactured by PT. Aventis Pharma, Indonesia.

DETAILED DESCRIPTION:
Twenty four healty volunteers were given a single dose of Furosemide 40 mg Tablet or Lasix® 40 mg Tablet with 240 mL of water beneath fasting condition. Then the blood samples for Furosemide were drawn and analyzed using UPLC. All subjects sample plasma were analyzed for pharmacokinetic evaluation

ELIGIBILITY:
Inclusion Criteria:

* have read the subject information and signed informed consent documents
* age 18 - 55 years
* body mass index between 18-25 kg/m2
* have a normal electrocardiogram
* blood pressure within normal range (systolic 90-120 mmHg and diastolic 60-80 mmHg)
* heart rate within normal range (60-100 bpm)
* with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening
* acceptance to use protection (condom) during intercourse with their spouse throughout the study

Exclusion Criteria:

* those who are pregnant and/or nursing women
* those with a history of hypersensitivity to furosemide, or other diuretics or other ingredients in the drugs or a history of serious allergic reaction to any drug, a significant allergic disease, or allergic reaction
* those with a history or presence of medical condition which might significantly influence the pharmacokinetic of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.
* those with a history or presence of any coagulation disorder or clinically significant hematology abnormalities
* those who are using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day
* those who have participated in any clinical study within 3 months prior to the study (< 90 days)
* those who have donated or lost 300 ml (or more) of blood within 3 months prior to the study
* those who smoke more than 10 cigarettes a day
* those who are positive to HIV, HBsAg, and HCV tests (to be kept confidential)
* those with a history of drug or alcohol abuse within 12 months prior to screening for this study
* those who are unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans D Suyatna, Principal Investigator — PT Pharma Metric Labs; I Gusti Putu Bagus Diana Virgo, Study Director — PT Pharma Metric Labs
Locations (1):
- PT Pharma Metric Labs, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Result] Chow SC. Bioavailability and Bioequivalence in Drug Development. Wiley Interdiscip Rev Comput Stat. 2014;6(4):304-312. doi: 10.1002/wics.1310. PMID 25215170
- [Result] Oh SW, Han SY. Loop Diuretics in Clinical Practice. Electrolyte Blood Press. 2015 Jun;13(1):17-21. doi: 10.5049/EBP.2015.13.1.17. Epub 2015 Jun 30. PMID 26240596
- [Result] Najib N, Idkaidek N, Beshtawi M, Bader M, Admour I, Alam SM, Zaman Q, Dham R. Bioequivalence evaluation of two brands of furosemide 40 mg tablets (Salurin and Lasix) in healthy human volunteers. Biopharm Drug Dispos. 2003 Sep;24(6):245-9. doi: 10.1002/bdd.361. PMID 12973821
- [Result] Shankar SS, Brater DC. Loop diuretics: from the Na-K-2Cl transporter to clinical use. Am J Physiol Renal Physiol. 2003 Jan;284(1):F11-21. doi: 10.1152/ajprenal.00119.2002. PMID 12473535
- [Result] Brater DC. Diuretic therapy. N Engl J Med. 1998 Aug 6;339(6):387-95. doi: 10.1056/NEJM199808063390607. No abstract available. PMID 9691107
- [Result] Sica DA. Diuretic use in renal disease. Nat Rev Nephrol. 2011 Dec 20;8(2):100-9. doi: 10.1038/nrneph.2011.175. PMID 22183505
- [Result] Ponto LL, Schoenwald RD. Furosemide (frusemide). A pharmacokinetic/pharmacodynamic review (Part I). Clin Pharmacokinet. 1990 May;18(5):381-408. doi: 10.2165/00003088-199018050-00004. PMID 2185908
- [Result] Midha KK, McKay G. Bioequivalence; its history, practice, and future. AAPS J. 2009 Dec;11(4):664-70. doi: 10.1208/s12248-009-9142-z. Epub 2009 Oct 6. No abstract available. PMID 19806461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 healthy volunteers were recruited from one research
Groups:
- Test Drug First, Then Reference Drug: New (test) Furosemide 40 mg tablet with 240 mL of water as a single oral dose in the first intervention period, and marketed (reference) Lasix® 40 mg tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period).
- Reference Drug First, Then Test Drug: Marketed (reference) Lasix® 40 mg tablet with 240 mL of water as a single oral dose in the first intervention period, and new (test) Furosemide 40 mg tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period)
Period: 1st Intervention
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Periods >= One Week
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: 2nd Intervention
Arm/Group | Test Drug First, Then Reference Drug | Reference Drug First, Then Test Drug
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 24 healthy volunteers
Groups:
- Total Number of Participants: All volunteers received Furosemide 40 mg tablet with 240 mL of water new and marketed)
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio of Maximum Concentration
Description: The ratio between test drug and reference drug
Time Frame: before dosing (0 h) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after drug administration
Measure: Geometric Mean (90% Confidence Interval); unit: percentage
Groups:
- Furosemide 40 mg Tablet: All volunteers received Furosemide 40 mg tablet with 240 mL of water (new and marketed drug)
Arm/Group | Furosemide 40 mg Tablet
Number analyzed (Participants) | 24
percentage | 104.51 [90.81 to 120.29]

2. Primary Outcome: Geometric Mean Ratio of Area Under Curve
Description: The ratio between test drug and reference drug
Time Frame: before dosing (0 h) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after drug administration
Measure: Geometric Mean (90% Confidence Interval); unit: percentage
Arm/Group | Furosemide 40 mg Tablet
Number analyzed (Participants) | 24
percentage | 101.79 [95.08 to 108.98]

3. Secondary Outcome: Pharmacokinetics Parameter
Description: Maximum plasma concentration
Time Frame: before dosing (0 h) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Furosemide 40 mg Tablet: volunteers received Furosemide 40 mg tablet with 240 mL of water (test drug)
- Lasix® 40 mg Tablet: volunteers received Lasix® 40 mg tablet with 240 mL of water (marketed drug)
Arm/Group | Furosemide 40 mg Tablet | Lasix® 40 mg Tablet
Number analyzed (Participants) | 24 | 24
ng/mL | 1893.09 (479.62) | 1907.32 (707.72)

4. Secondary Outcome: Pharmacokinetics Parameter
Description: Area Under Curve from 0 to 24 hours
Time Frame: before dosing (0 h) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Furosemide 40 mg Tablet | Lasix® 40 mg Tablet
Number analyzed (Participants) | 24 | 24
ng*h/mL | 4938.79 (1110.92) | 4921.94 (1279.14)

ADVERSE EVENTS:
Time Frame: before dosing (0 h) and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours
Description: [Not Specified]
Arm/Group | Furosemide 40 mg Tablet | Lasix® 40 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 5/24 | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide 40 mg Tablet (N=24) | Lasix® 40 mg Tablet (N=24)
Headache (Nervous system disorders) | 3 (5) | 2 (5)
Polyuria (Gastrointestinal disorders) | 1 (3) | 2 (3)
Frequent urination (Gastrointestinal disorders) | 2 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04982874/Prot_SAP_000.pdf